CLINICAL TRIAL: NCT01040221
Title: Trichuris Suis Ova in Autism Spectrum Disorders
Acronym: TSO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Simons Foundation (Other)
Responsible Party: Principal Investigator, Eric Hollander, Clinical Professor, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-11-384
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Autism
Keywords: Autism, Autism Spectrum Disorder; ASD; Trichuris Suis Ova; TSO; Treatment; Clinical Trial
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trichuris Suis Ova (TSO) (Experimental): the eggs of intestinal helminthes (trichuris suis ova) administered as 2500 ova doses every two weeks.
  Interventions: Drug: Trichuris Suis Ova
- Placebo (Placebo Comparator): placebo dosage received every two weeks.
  Interventions: Drug: Trichuris Suis Ova

INTERVENTIONS:
Drug: Trichuris Suis Ova — TSO will be administered in vials prepared by Coronado Biosciences. Vials will be diluted with a commercial drink and given to subjects to ingest. Subjects will receive a dose of 2500 ova every two weeks for 12 weeks.

SUMMARY:
The purpose of this study is to determine whether Trichuris Suis Ova (TSO) is safe and effective in treating adults with autism spectrum disorder

DETAILED DESCRIPTION:
Autism is a pervasive developmental disorder affecting social, communicative, and compulsive/repetitive behaviors. It is also frequently accompanied by aggression, self-injury, and irritability, making care for these individuals a significant challenge for families or institutional settings. Currently risperidone is the only medication approved by the Food and Drug Administration (FDA) for irritability associated with autism, although not all patients respond to risperidone or are able to tolerate its side effects. As such, additional targeted treatments need to be explored in autism. Neuroimmune disturbance has been demonstrated in patients with autism (Ashwood et al., 2006; DelGuidice, 2003) and the presence of neuroinflammation may play a role in initiating or maintaining CNS dysfunction characteristic of the disorder (Pardo et al, 2005). Therefore, there is considerable interest in using immunomodulatory medications to address core and associated symptoms.

Trichuris suis ova (TSO) are the eggs of intestinal helminthes which induce Th2 cytokine release and nonspecifically downregulate Th1 responsiveness (Summers et al., 2003). Treatment with TSO has been shown to have a beneficial effect in autoimmune inflammatory bowel disease (Summers et al, 2003; Summers et al., 2005a; Summers et al., 2005b) and anecdotal reports from patients with autism have demonstrated that TSO may be effective in reducing repetitive behaviors, aggression, self-injury, and impulsivity.

To date, many medications have been used in individuals with autism and the history of psychopharmacology of autism is notable for the exaggerated benefit of a variety of treatments. To date, most medication studies in the field have been open-label without use of a placebo control and without systematic behavioral assessments. The current practice of prescribing medications to patients with autism without scientifically demonstrated efficacy underscores the necessity for methodologically rigorous studies to be conducted.

We propose a double blind placebo-controlled crossover trial of TSO, where subjects would be randomized to receive placebo or TSO for 12 weeks, with a 4 week washout and then 12 weeks of the the treatment not yet received. To assess the effect on social cognition, repetitive behaviors, aggression and irritability, and global functioning in adults with autism spectrum disorder. The objectives of the proposed study are to develop an innovative treatment approach to autism by 1) assessing the safety and efficacy of TSO treatment using behavioral and laboratory outcome measures; 2) determining whether this treatment has sufficient promise to warrant consideration of a larger, multi-centered, placebo-controlled clinical trial; 3) conducting secondary analyses to explore the relationship between clinical features, immune mechanisms, and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35, inclusive, at the time of consent
2. Outpatient
3. Meet criteria for the diagnosis of Autism Spectrum Disorder according to the DSM-IV-TR, and supported by the ADOS or ADI-R.
4. Have an IQ of 70 or greater
5. Participants who are taking other medications prior to enrollment must be on a stable dose of concomitant medication, including psychotropic, anticonvulsant, or sleep aid for at least 3 months prior to baseline ratings
6. Be judged reliable for medication compliance and agree to keep appointments for study contacts and tests as outlined in the protocol (both subjects and guardians)
7. Have a personal or family history of allergies.

Exclusion Criteria:

1. History of Bipolar disorder or Psychotic Disorders (e.g. schizophrenia or schizoaffective disorders).
2. Previous diagnosis of Rett's Disorder or Childhood Disintegrative Disorder
3. Uncontrolled seizure disorders (seizures within the past 6 months)
4. Pregnant or breast feeding at screening, or at any time during the study
5. Chronic medical illness that would interfere with or contraindicate participation in the study, or clinically significant abnormalities in baseline laboratory testing or physical exam.
6. Treatment in the last 12 weeks with cyclosporine, methotrexate, infliximab or immunomodulatory agents
7. Treatment in the last 2 weeks with antibiotics, antifungal or antiparasitic medications
8. Presence of any organic or systemic disease or need for a therapeutic intervention, which would confound the interpretation of results.
9. History of previous treatment with Trichuris Suis Ova (TSO).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS): to measure repetitive behaviors | baseline, 2, 4, 6, 8, 10, 12, 14, 16 weeks
Aberrant Behavior Checklist (ABC): to measure aggression and irritability | baseline, 2, 4, 6, 8, 10, 12, 14, 16 weeks
Clinical Global Impression - Improvement (CGI-I): to measure global functioning | baseline, 2, 4, 6, 8, 10, 12, 14, 16 weeks

SECONDARY OUTCOMES:
Repetitive Behavior Scale-Revised. | baseline, 2, 4, 6, 8, 10, 12, 14, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Hollander E, Uzunova G, Taylor BP, Noone R, Racine E, Doernberg E, Freeman K, Ferretti CJ. Randomized crossover feasibility trial of helminthic Trichuris suis ova versus placebo for repetitive behaviors in adult autism spectrum disorder. World J Biol Psychiatry. 2020 Apr;21(4):291-299. doi: 10.1080/15622975.2018.1523561. Epub 2018 Nov 16. PMID 30230399